CLINICAL TRIAL: NCT04096079
Title: Post-ROSC Electrocardiogram After Cardiac arrEst
Acronym: PEACE
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Nicosia General Hospital (Other); Cardiocentro Ticino (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Simone Savastano, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PEACE Study
Record Dates: First submitted 2019-09-14; First posted 2019-09-19 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Infarction, Myocardial
Keywords: Out-Of-Hospital Cardiac Arrest, STEMI, coronary angiography, post-ROSC ECG
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA patients: Patients who suffered an out-of-hospital cardiac arrest between 2015 and 2018 in Province of Pavia (Italy), Ticino Region (Switzerland), Wien area (Austria) and Nicosia area (Cyprus) who underwent a coronary angiography.

SUMMARY:
PEACE study retrospectively evaluate patients who suffered an out-hospital cardiac arrest (OHCA) and who underwent a coronary angiography, enrolled in the registry of the Province of Pavia (Italy), Ticino Region (Switzerland), Wien region (Austria) and Nicosia area (Cyprus) to comprehend the best timing for post-ROSC ECG acquisition in order to reduce the number of false positive and to select the best candidates for emergency coronary angiography.

DETAILED DESCRIPTION:
Twelve leads electrocardiogram (ECG) represents an essential step of the diagnostic workflow after ROSC as stated by both the European and the American guidelines. Actually about 80% of patients showing an ST segment elevation after return of spontaneous circulation (ROSC) have a coronary lesion documented by coronary angiography. In those patients, early coronary angiography has been shown to improve survival with good neurologic outcome. More controversial is the scene for patients without an ST segment elevation. Even in the absence of ST segment elevation an acute coronary syndrome can be at the basis of cardiac arrest. However, the prognostic role of early coronary angiography in such patients is still a matter of debate. In 2014 a consensus document by the European Association for Percutaneous Cardiovascular Interventions (EAPCI) recommended elevation to consider early coronary angiography only in the case of hemodynamic instability or of recurrent ventricular arrhythmias for patients without ST segment as in the case of NSTEMI patients without cardiac arrest. At the light of these considerations the correct diagnosis of ST segment elevation is of pivotal importance for the right treatment in the right time and in the right hospital for this type of patients. Moreover, during cardiac arrest and during resuscitation the heart is suffering of ischemia deriving both from a coronary occlusion if present and from low systemic perfusion. Post-ROSC ECG could reflect both these types of ischemia, so the ST elevation could be not specific for a coronary occlusion. However, some time after ROSC, in case of absence of a coronary occlusion, the heart perfusion should improve, the ischemia should decrease and the ST segment elevation should regress. Nevertheless, current guidelines do not provide any indication about the best timing for ECG acquisition after ROSC. We believe that address this issue could be important in order to correctly discriminate the appropriate candidate for emergency coronary angiography in the post-ROSC phase of a cardiac arrest.

A preliminary analysis performed on a population of patients suffering an OHCA in the Province of Pavia supported this hypothesis. It was pointed out that early detection of ST segment elevation, within ten minutes from ROSC, was associated to a high number of false positives that is to say patients without an identifiable coronary culprit lesion. ST segment elevation was found to be an independent predictor of coronary angioplasty only if detected after ten minutes from ROSC.

The PEACE study aimed to confirm our preliminary results on a larger and multicentric sample of post ROSC patients.

ELIGIBILITY:
Inclusion Criteria:

* All the patients older than 18 years old resuscitated from an out-of-hospital cardiac arrest with an available post-ROSC twelve leads ECG who underwent to a coronary angiography during hospital stay.

Exclusion Criteria:

* From the present study are excluded all the patients with a non-medical aetiology of the cardiac arrest (trauma, drowning, electrocution, drug or abuse substance overdose, asphyxia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OHCA patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint - PCI | Up to 14 days after OHCA (hospital discharge)
  To assess the number of patients requiring a coronary angioplasty in the presence of ST segment elevation according to the ROSC-ECG time
Primary endpoint - Time | Up to 14 days after OHCA (hospital discharge)
  To identify the ROSC-ECG time associated to the lowest rate of false positive

SECONDARY OUTCOMES:
Secondary outcome - PCI in STEMI patients | Up to 14 days after OHCA (hospital discharge)
  to assess the number of patients requiring a coronary angioplasty in the absence of ST segment elevation
Secondary outcome - PCI in BBB patients | Up to 14 days after OHCA (hospital discharge)
  to assess the number of patients requiring a coronary angioplasty in the presence of left or right bundle branch block